CLINICAL TRIAL: NCT03654391
Title: Study of Obesity Control by Astragalus and Notoginseng Extrats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, School of Health Diet and Industry Managment, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS16098
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: Astragalus and Notoginseng extrats; Body weight; BMI; Triglyceride; obese
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InnoSlim (Active Comparator): Subjects ingested 2 capsules InnoSlim® (Experimental group) in the morning and 3 capsules in the evening (5 capsules/d) for 12 weeks of a stage.
  Interventions: Dietary Supplement: InnoSlim
- Placebo (Placebo Comparator): Subjects ingested 2 capsules placebo (Control group) in the morning and 3 capsules in the evening (5 capsules/d) for 12 weeks of a stage.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: InnoSlim — Subjects ingested 2 capsules (Experimental group) in the morning and 3 capsules in the evening (5 capsules/d) for 12 weeks of a stage. Anthropometric measurements such as body weight, body fat, waistline, hipline, blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST and ALT were measured every six weeks.
  Other Names: Astragalus and Notoginseng extrats
  Arms: InnoSlim
Dietary Supplement: Placebo — Subjects ingested 2 capsules placebo in the morning and 3 capsules in the evening (5 capsules/d) for 12 weeks of a stage. Anthropometric measurements such as body weight, body fat, waistline, hipline, blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST and ALT were measured every six weeks.
  Arms: Placebo

SUMMARY:
The effects of the Astragalus and Notoginseng extrats on obesity control was demonstrated in a randomized double-blind, and crossover human trial.

DETAILED DESCRIPTION:
Obesity refers to the body due to physiological or biochemical function of the change caused by excessive accumulation of body fat, resulting in weight gain. Hence, the aim of this study was to evaluate the effects of the Astragalus and Notoginseng extrats on obesity control by a randomized double-blind and crossover human trial. Subjects with simple obesity (body mass index (BMI) ≥ 27 or body fat ≥ 30%) ingested 5 extrats (n = 19) capsules or placebo (n = 19) perday for 12 weeks of a stage. Anthropometric measurements (body weight, body fat, blood pressure) and blood biochemical markers including fasting blood glucose (FBG), albumin, total cholesterol (TC), triglyceride (TG), HDL-C, LDL-C, creatinine (Cr), blood urea nitrogen (BUN), AST, ALT were examined every six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 27 or body fat ≥ 30%;
* No history of serious diseases associated with heart, liver, kidney, endocrine systems or other organs;
* No drugs consumption.

Exclusion Criteria:

* BMI >35;
* Alcoholic;
* US-controlled diabetics;
* Stoke in past one year;
* High blood pressure;
* Mental diseases or melancholia;
* Pregency or breast-feeding a child.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The changes of body weight and BMI of the subjects. | 12 weeks
  values change of body weight and BMI between before to after 12 weeks

SECONDARY OUTCOMES:
The changes of triglyceride (TG) of the subjects | 12 weeks
  values change of triglyceride (TG) between before to after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: irb@csh.org.tw Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University

REFERENCES:
- [Result] Chang W.L. et al. The inhibitory effect of ginse¬noside Rg1 on glucose and lipid production in human HepG2 cells. Adaptive Medicine. 2013, 5(4), 181-188.
- [Result] Chang TC, Huang SF, Yang TC, Chan FN, Lin HC, Chang WL. Effect of ginsenosides on glucose uptake in human Caco-2 cells is mediated through altered Na+/glucose cotransporter 1 expression. J Agric Food Chem. 2007 Mar 7;55(5):1993-8. doi: 10.1021/jf062714k. Epub 2007 Feb 2. PMID 17269785
- [Result] Wang CW, Su SC, Huang SF, Huang YC, Chan FN, Kuo YH, Hung MW, Lin HC, Chang WL, Chang TC. An Essential Role of cAMP Response Element Binding Protein in Ginsenoside Rg1-Mediated Inhibition of Na+/Glucose Cotransporter 1 Gene Expression. Mol Pharmacol. 2015 Dec;88(6):1072-83. doi: 10.1124/mol.114.097352. Epub 2015 Oct 1. PMID 26429938